CLINICAL TRIAL: NCT03063710
Title: Olaparib Expanded Access Program for BRCA Mutated Platinum Sensitive Relapsed High Grade Epithelial Ovarian Cancer Patients
Brief Title: Olaparib Expanded Access Program for BRCA Mutated Platinum Sensitive Relapsed High Grade Epithelial Ovarian Cancer Patients in Japan
Status: No longer available | Type: Expanded Access
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D0816L00006
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: PSR Ovarian Cancer With a BRCA Mutation
MeSH Terms: interventions — olaparib

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: olaparib — Initial dose is 300mg twice daily. Study treatment can be dose reduced to 250 mg bd as a first step and to 200 mg bd as a second step. There is no maximum duration for taking study treatment. Patients may continue to receive study treatment until disease progression as assessed by the investigator according to local standard clinical practice or any other discontinuation criteria.

SUMMARY:
This is a single-arm, open label, expanded access program to provide access to olaparib tablets for relapsed high-grade epithelial ovarian cancer patients (including patients with primary peritoneal and / or fallopian tube cancer) with BRCA mutations (documented mutation in BRCA1 or BRCA2 that is predicted to be deleterious or suspected deleterious [known or predicted to be detrimental/lead to loss of function]) who have responded following platinum based chemotherapy.

Patients may continue to receive study treatment until disease progression as assessed by the investigator according to local standard clinical practice or any other discontinuation criteria are met.

DETAILED DESCRIPTION:
Primary Objective:

To provide expanded access to olaparib tablets for use as maintenance monotherapy in BRCA mutated platinum sensitive relapsed (PSR) high grade epithelial ovarian cancer patients who are in complete or partial response following platinum based chemotherapy.

Secondary Objective:

Not applicable

Safety Objective:

To collect the individual safety data of olaparib maintenance monotherapy in BRCA mutated PSR high grade epithelial ovarian cancer patients who are in complete or partial response following platinum based chemotherapy.

When the number of enrolled patients is not enough (<5 patients), only listings of safety data will be prepared. On the other hand, if the number is sufficient (>=5 patients), summaries of safety data will be prepared using descriptive statistics.

Target subject population Patients with PSR high-grade epithelial ovarian cancer with a BRCA mutation (this includes any patients with primary peritoneal and / or fallopian tube cancer). At enrollment, patients will be in complete or partial response following completion (a minimum of 4 treatment cycles) of platinum-based chemotherapy.

Patients must have completed at least 2 previous lines of platinum-based therapy (e.g., carboplatin or cisplatin) before entry to the study and must be considered platinum sensitive after the penultimate platinum-based chemotherapy. Platinum sensitive in this study is defined as disease progression greater than 6 months after completion (last dose) of the penultimate platinum chemotherapy.

Patients must not have received bevacizumab during the chemotherapy course immediately prior to entry. Cytoreductive surgery prior to the end of the last chemotherapy regimen is allowed as long as it is completed before the end of the chemotherapy regimen.

Patients known to have BRCA mutation/s from germline (i.e., blood) or a tumour specimen, prior to provision of informed consent can enter the study based on this result. The result must be made available to AstraZeneca. Patients that have a BRCA mutation identified can enter the study provided that all such testing has been undertaken in appropriately accredited laboratories.

Duration of treatment Patients may continue to receive study treatment until disease progression as assessed by the investigator according to local standard clinical practice or any other discontinuation criteria are met.

Investigational product, dosage and mode of administration Olaparib is available as a film-coated tablet containing 150 mg or 100 mg of olaparib. Patients will be administered study treatment orally at a dose of 300 mg twice daily. The planned dose of 300 mg twice daily will be made up of two x 150 mg tablets twice daily with 100 mg tablets used to manage dose reductions.

Statistical methods Approximately 10 patients will be allowed to enter the expanded access program. No formal analysis will be performed on any data obtained. However all safety data will be summarised and tabulated for regulatory purposes only, if the number of enrolled patients is sufficient (>= 5 patients). On the other hand, if the number of patients is small (<5 patients), only listings of safety data will be prepared.

If the number of enrolled patients is sufficient, data summaries will be prepared based on the Safety Analysis Set, which will consist of patients who have received at least one dose of olaparib and have at least one post baseline safety assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Patients must be a permanent resident in Japan and ≥ 18 years of age. For patients aged under 20 years, written informed consent should be obtained both from the patient and his/her legal representative.
3. Female patients with histologically diagnosed high grade epithelial ovarian cancer
4. Documented mutation in BRCA1 or BRCA2 that is predicted to be deleterious or suspected deleterious from germline or a tumour specimen, prior to provision of informed consent
5. Patients who have received at least 2 previous lines of platinum containing therapy prior to assignment to the study

   1. For the chemotherapy course prior to assignment to the study (except (b)):

      * Treatment must have contained a platinum agent
      * Patient defined as platinum sensitive after this treatment; defined as disease progression greater than 6 months after completion of their last dose of platinum chemotherapy
      * Maintenance treatment is allowed at the end of the penultimate platinum regimen, including bevacizumab
   2. For the last chemotherapy course immediately prior to assignment to the study

      * Patients must be, in the opinion of the investigator as per local standard clinical practice, in response or may have no evidence of disease, and no evidence of a rising CA-125, as defined below, following completion of this chemotherapy course
      * Patient must have received a platinum based chemotherapy regimen and have received at least 4 cycles of treatment
      * Patients must not have received bevacizumab during this course of treatment
      * Patients must not have received any investigational agent during this course of treatment
      * Patients must be assigned within 8 weeks of their last dose of chemotherapy
6. Pre-treatment CA-125 measurements must meet criterion specified below:

   * If the first value is within ULN the patient is eligible to be randomised and a second sample is not required
   * If the first value is greater than ULN a second assessment must be performed at least 7 days after the 1st. If the second assessment is ≥ 15% more than the first the patient is not eligible
7. Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment, as defined below:

   * Haemoglobin ≥ 10.0 g/dL with no blood transfusions in the past 28 days
   * ANC ≥ 1.5 x 109/L
   * Platelet count ≥ 100 x 109/L
   * Total bilirubin ≤ 1.5 x institutional upper limit of normal
   * AST/ALT ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case they must be ≤ 5x ULN
   * Patients must have creatinine clearance estimated using the Cockcroft-Gault equation of ≥ 51 mL/min:
8. ECOG performance status 0-1
9. Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test

   Postmenopausal is defined as:
   * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
   * LH and FSH levels in the post menopausal range for women under 50
   * radiation-induced oophorectomy with last menses >1 year ago
   * chemotherapy-induced menopause with >1 year interval since last menses
   * or surgical sterilisation
10. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations

Exclusion Criteria:

1. BRCA1 and/or BRCA2 mutations that are considered to be non detrimental
2. Patients who have had drainage of their ascites during the final 2 cycles of their last chemotherapy regimen prior to assignment to the study
3. Previous assignment to the present study
4. Participation in another clinical study with an investigational product during the chemotherapy course immediately prior to assignment
5. Any previous treatment with a PARP inhibitor, including olaparib
6. Patients with a known hypersensitivity to olaparib or any of the excipients of the product
7. Resting ECG with QTc > 470 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome
8. Patients receiving any systemic chemotherapy or radiotherapy within 3 weeks prior to study treatment.
9. Concomitant use of known strong CYP3A inhibitors or moderate CYP3A inhibitors. The required washout period prior to starting study treatment is 2 weeks.
10. Concomitant use of known strong or moderate CYP3A inducers. The required washout period prior to starting study treatment is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
11. Persistent toxicities (>CTCAE grade 2) caused by previous cancer therapy, excluding alopecia
12. Patients with MDS/AML or with features suggestive of MDS/AML.
13. Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days
14. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery
15. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on HRCT scan or any psychiatric disorder that prohibits obtaining informed consent.
16. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication
17. Breast feeding women
18. Immunocompromised patients
19. Patients with known active hepatitis due to risk of transmitting the infection through blood or other body fluids
20. Previous allogenic bone marrow transplant or dUCBT
21. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Research Site, Akashi-shi, Hyōgo
  - Research Site, Chuo-ku, Tokyo